CLINICAL TRIAL: NCT03466983
Title: A Randomized, Double-blinded, Comparative Trial Comparing the Incidence of Hypophosphatemia in Relation to Repeated Treatment Courses of Iron Isomaltoside and Ferric Carboxymaltose in Subjects With Iron Deficiency Anaemia Due to Inflammatory Bowel Disease
Brief Title: A Trial Comparing the Incidence of Hypophosphatemia in Relation to Treatment With Iron Isomaltoside and Ferric Carboxymaltose in Subjects With Iron Deficiency Anaemia Due to Inflammatory Bowel Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pharmacosmos A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P-Monofer-IBD-03
Record Dates: First submitted 2018-03-06; First posted 2018-03-15 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: IBD
MeSH Terms: interventions — iron isomaltoside 1000; ferric carboxymaltose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iron Isomaltoside (Experimental): Iron Isomaltoside (Monofer) administered IV
  Interventions: Drug: Iron Isomaltoside
- Ferric Carboxymaltose (Active Comparator): Ferric Carboxymaltose (Injectafer) administered IV
  Interventions: Drug: Ferric Carboxymaltose

INTERVENTIONS:
Drug: Iron Isomaltoside — administered IV
  Other Names: Monofer
  Arms: Iron Isomaltoside
Drug: Ferric Carboxymaltose — administered IV
  Other Names: Ferinject
  Arms: Ferric Carboxymaltose

SUMMARY:
Treatment with iron isomaltoside and ferric carboxymaltose in subjects with iron deficiency anaemia due to inflammatory bowel disease and comparison of the incidence of hypophosphatemia

DETAILED DESCRIPTION:
Existing IV iron complexes differ in relation to the compounds capability to induce unintended hypophosphatemia to a degree defined as medical significant.

This trial is designed evaluate the effect of IV iron isomaltoside compared to IV ferric carboxymaltose on phosphate in subjects with IDA due to inflammatory bowel disease .

ELIGIBILITY:
Inclusion Criteria include:

* Men or women ≥ 18 years
* Subjects diagnosed with IBD
* Hb < 13 g/dL
* Body weight ≥ 50 kg
* S-ferritin <100 ng/mL
* eGFR ≥ 65 mL/min/1.73 m2
* S-phosphate > 2.5 mg/dL
* Oral iron preparations are ineffective or cannot be used or where there is a clinical need to de-liver iron rapidly
* Willingness to participate and signing the Informed Consent Form (ICF)

Exclusion Criteria include:

* Anaemia predominantly caused by factors other than IDA according to Investigator's judgment
* Hb ≥ 10 g/dL and body weight < 70 kg
* Hemochromatosis or other iron storage disorders
* Known hypersensitivity reaction to any component of iron isomaltoside or ferric carboxymaltose
* Previous serious hypersensitivity reactions to any IV iron compounds
* Treatment with IV iron within the last 30 days prior to screening
* Treatment with erythropoietin or erythropoietin-stimulation agents, red blood cell transfusion, radiotherapy, and/or chemotherapy within the last 30 days prior to screening
* Received an investigational drug within the last 30 days prior to screening
* Planned surgical procedure within the trial period
* hepatic enzymes > 3 times upper limit of normal
* Surgery under general anaesthesia within the last 30 days prior to screening
* Any non-viral infection within the last 30 days prior to screening
* Alcohol or drug abuse within the past 6 months
* Untreated hyperparathyroidism
* Kidney transplantation
* Conditions that interfere with the subject's ability to understand the requirements of the trial and/or presumable non-compliance
* Any other laboratory abnormality, medical condition, or psychiatric disorders which, in the opinion of the Investigator, will put the subject's disease management at risk or may result in the subject being unable to comply with the trial requirements
* Pregnant or nursing women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2018-05-23 (Actual); Primary Completion 2020-05-25 (Actual); Study Completion 2020-05-25 (Actual)

PRIMARY OUTCOMES:
Incidence of hypophosphatemia | any time from baseline to day 35
  s-phosphate < 2 mg/dL

SECONDARY OUTCOMES:
Incidence of hypophosphatemia | any time from baseline to week 10
  s-phosphate < 2 mg/dL
Incidence of s-phosphate < 1.0 mg/dL | any time from baseline to day 35
  s-phosphate < 1.0 mg/dL
Time with hypophosphatemia | number of days any time from baseline to week 10
  time with s-phosphate < 2.0 mg/dL

CONTACTS AND LOCATIONS:
Locations (1):
- Pharmacosmos Investigational Site, Silkeborg, Denmark

REFERENCES:
- [Derived] Bjorner JB, Kennedy N, Lindgren S, Pollock RF. Hypophosphatemia attenuates improvements in vitality after intravenous iron treatment in patients with inflammatory bowel disease. Qual Life Res. 2024 Aug;33(8):2285-2294. doi: 10.1007/s11136-024-03642-y. Epub 2024 Jun 14. PMID 38874697